CLINICAL TRIAL: NCT01320891
Title: Effects of Different Strategy of Fluids Administration on Acid/Base Disorders and Inflammatory Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Principal Investigator, Carlo Alberto Volta, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-I-H-0909
Record Dates: First submitted 2011-03-08; First posted 2011-03-23 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Large Bowel Cancer
Keywords: general anaesthesia for major abdominal surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — sterofundin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- balanced (Experimental): arm in which the subjects received only balanced solutions
  Interventions: Behavioral: balanced solutions
- not balanced (Experimental): arm in which the subjects received only not balanced solutions that means only normal saline and colloid dissolved in normal saline
  Interventions: Behavioral: not balanced

INTERVENTIONS:
Behavioral: balanced solutions — during the general anaesthesia until 8 o'clock of the day after the operation the subject will receive only balanced fluids that means balanced crystalloid and colloids dissolved in balanced solution. 12 ml /Kg/h during operation time. ratio 3:1 between crystalloid and colloid.
  Other Names: sterofundin, tetraspan
  Arms: balanced
Behavioral: not balanced — during the operation time until the 8 o'clock of the day after the operation, the subjects will receive only normal saline and colloid dissolved in normal saline.
  Other Names: Normal saline, Amidolite
  Arms: not balanced

SUMMARY:
Aim of the study is to ascertain whether a different strategy of fluids administration can be responsible of differences in terms of acid/base disorders (Stewart approach), pro-inflammatory and inflammatory mediators. Hence two groups of patients will be treated either with not-balanced solutions (Normal Saline) or balanced solutions

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of large bowel cancer
* Age > 18 years old

Exclusion Criteria:

Emergency surgery for bowel punch or intestinal occlusion

* Massive bleeding
* Therapy with corticosteroid or nonsteroid antiinflammatory substances
* Renal insufficiency (serum creatinine > 200 micromol /l)
* Cardiac insufficiency (NYHA III-IV)
* Altered liver function (ALT > 40 U/l AST >40 U/l)
* Preoperative anaemia ( Hb < 10 g/dl )
* Allergy to hydrossietilic starches
* Patient rejection to share the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
acid/base disorder | T0: anaesthesia induction (control value) T1: end of surgery T2: 1h after the end of surgery T3: 24h after the beginning of surgery
  the investigators assess difference in acid base disorders between the two groups measuring emogas analyses data and blood electrolites levels at the same time (two days)

SECONDARY OUTCOMES:
pro/antiinflammatory cytokine | T0: anaesthesia induction (control value) T1:end of surgery T2: 1h after the end of surgery T3: 24h after the beginning of surgery
  -MMP-9 total and active, TIMP-1, IL-6, IL-8, IL-10, mieloperossidasis, ROS, MCP-3 will be measured during the observation period. (two days)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo A Volta, Professor, Study Chair — Ferrara Univesity
Locations (1):
- S.Anna Universitary Hospital, Ferrara, Italy

REFERENCES:
- [Derived] Volta CA, Trentini A, Farabegoli L, Manfrinato MC, Alvisi V, Dallocchio F, Marangoni E, Alvisi R, Bellini T. Effects of two different strategies of fluid administration on inflammatory mediators, plasma electrolytes and acid/base disorders in patients undergoing major abdominal surgery: a randomized double blind study. J Inflamm (Lond). 2013 Sep 24;10(1):29. doi: 10.1186/1476-9255-10-29. PMID 24059479